CLINICAL TRIAL: NCT06832891
Title: A Survey of Patient Preferences on Empathetic Communication in Outpatient Palliative Care
Brief Title: Patient Preferences in Empathetic Communication by AI vs Human Authorship
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 24-010821
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Preference, Patient
Keywords: AI
MeSH Terms: conditions — Patient Preference | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survey Group - Blinded: Participants will be blinded to origin of survey statements
  Interventions: Other: Survey
- Survey Group - Unblinded: Participants will be informed of origin of survey statements
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Patients complete survey

SUMMARY:
This study aims to evaluate whether patients have different preference patterns for empathetic communication through AI vs human-being when knowledge of authorship is known vs blinded.

DETAILED DESCRIPTION:
Hypothesis:

Patients will express increased preference for human-generated empathetic communication vs AI-generated empathetic communication when they are made aware of authorship vs when blinded to it.

Aims, purpose, or objectives:

Evaluate if patients have different preference patterns for empathetic communication through AI vs human-being when knowledge of authorship is known vs blinded

Background:

Artificial intelligence (AI) is rapidly gaining a foothold in the healthcare industry. AI's role in healthcare can largely be divided into two sets of tasks: Those which involve direct interaction with patients and those which do not. Many tasks which do not directly interact with patients, such as monitoring and resupplying medications, delivering goods across a hospital, and analyzing practice trends and outcomes are highly likely to benefit from the efficiency, cost-savings, and consistency AI can provide. Tasks involving direct patient interaction are considerably more controversial. Understanding of how patients will respond to AI communication remains quite limited which is concerning considering the rapid expansion of AI into the healthcare space. A logical first step to investigate is to see if patients react to AI communication when they are blinded to it vs when authorship is known. This concept has previously been tested in other industries such as business and the law, but patient communication preference in healthcare has been little studied, especially in palliative care. It is the aim of this study to investigate this.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 being seen in palliative care clinic who have already established care and with diagnosis of any malignancy

Exclusion Criteria:

* Inability to consent defined as: Acute mental status changes (delirium/encephalopathy), acute substance intoxication, intellectual disability, dementia, patient with active legal guardian
* Major psychiatric disorders including, but not limited to, bipolar disorder, psychotic disorders, active substance use disorder, and patients with active suicidal or homicidal thoughts.

  * NOTE: Patients with history of normal grieving reactions, major unipolar depressive disorder, posttraumatic stress disorder or generalized anxiety disorder would NOT be excluded.
* Inability to read in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 being seen in palliative care clinic who have already established care and with diagnosis of any malignancy
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2025-04-21 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Preference patterns for empathetic communication | Baseline
  Assessed by a brief survey: patients will be show two brief empathetic statements related to their serious illness diagnosis (Cancer), one generated by Artificial Intelligence (AI) and one generated by a human physician in palliative care who were both given the same writing instructions and generated their responses independently. Half of the surveys will label which statement is generated by human or AI unblinded group) and the other half will be blinded to statement authorship. Preference will be compared between the blinded and unblinded groups.

CONTACTS AND LOCATIONS:
Overall Officials: April Christensen, MD, MS, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials